CLINICAL TRIAL: NCT00951756
Title: Controlled Feeding Experiment of High and Low Fat Diet and Stool Microbiome Controlled Feeding Experiment of High and Low Fat Diet and Stool Microbiome Composition
Brief Title: Controlled Feeding Experiment
Acronym: CaFE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: James Lewis (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor-Investigator, James Lewis, Professor of Medicine and Epidemiology, University of Pennsylvania
Organization: University of Pennsylvania (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: DK83981; UH2DK083981 (NIH)
Record Dates: First submitted 2009-08-03; First posted 2009-08-04 (Estimated); Last update posted 2013-06-25 (Estimated); Status verified 2013-06

CONDITIONS: Effect of Diet on Microbiome Composition
Keywords: Dietary fat; Microbiome composition; Controlled feeding experiment
MeSH Terms: interventions — Diet, High-Fat

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- High Fat Low Fiber Diet (Other)
  Interventions: Other: High fat diet
- Low Fat High Fiber Diet (Other)
  Interventions: Other: High fat diet

INTERVENTIONS:
Other: High fat diet — High fat diet and low fat diet are composed of the same food, but the portion sizes are varied.

SUMMARY:
The purpose of this study is to determine the effect of dietary fat, in standard formulation, on the composition of the human microbiome in a prospective study of normal volunteers. Participants will be randomly assigned to either a high fat or low fat diet for 10 days. The gut microbiome will be phylotyped in fecal samples as well as in bacteria adherent to the colonic mucosa prior to, and during the course of the dietary interventions.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is capable of giving informed consent
2. Participant is age 18 to 40 years

Exclusion Criteria:

1. Diagnosis with Inflammatory bowel disease (IBD), celiac disease, or other chronic intestinal disorders.
2. Baseline bowel frequency less than every 2 days or greater than 3 times daily.
3. Current smoker.
4. Body Mass Index (BMI) <18.5 of >35.
5. Diabetes mellitus (DM)
6. Diagnosis with coronary artery disease, congestive heart failure, or prior myocardial infarction.
7. History of dyslipidemia or receiving treatment for hypercholesterolemia. This will be defined as a fasting LDL >160 mg/dL or a non-fasting total cholesterol >200 mg/dL or non-fasting HDL<40 mg/dl. Additionally, patients receiving drug therapy for hypercholesterolemia will be excluded.
8. Prior bowel resection surgery.
9. Contraindication to flexible sigmoidoscopy and biopsies. Patients with suppressed white blood count may be at increased risk of systemic infection following sigmoidoscopy with biopsies. As such, subjects with a white blood cell (WBC) count less than 3,500 or an absolute neutrophil count of less than 1,000 will be excluded. Patients with thrombocytopenia or with a coagulopathy may be at increased risk of bleeding complications after colonoscopic biopsies. As such, patients with a platelet count of less than 100,000 or an international normalized ratio (INR) greater than 1.2 will be excluded from the study.
10. Student or employee of any one of the investigators.
11. Pregnant women.
12. Use of antibiotics in the prior 6 months.
13. Use of antacids, non-steroidal anti-inflammatory drugs (NSAIDs), or dietary supplements in the preceding 2 weeks.
14. Use of any of the following medications in the 4 weeks prior to randomization: proton pump inhibitors (PPI), histamine receptor antagonists, narcotics, tricyclic antidepressants, anticholinergics (e.g., hyoscamine), metoclopramide, anti-diarrhea medications, laxatives.
15. HIV infection, AIDS, or other known conditions resulting in immunosuppression.
16. Allergies or intolerance to the components of the study diets.
17. Participant has experienced diarrhea within the two weeks prior to the first sigmoidoscopy. Diarrhea is defined as a change in bowel habits with an increased frequency or loose stools such that the stool could not be lifted with a fork.
18. Any condition that the investigator feels may limit the volunteer's ability to complete the study protocol.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2009-07; Primary Completion 2010-01 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
This is not an efficacy study. There is no pre-specified clinical endpoint for this study. Rather, the outcome is the composition of the gut microbiome. | 10 days

CONTACTS AND LOCATIONS:
Overall Officials: James D Lewis, MD, MSCE, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States